CLINICAL TRIAL: NCT00769574
Title: Assessment of New Biomarkers in the Management and Triage of Patients With Chest Pain and Suspicion of Non ST Elevation Acute Coronary Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-A00192-53
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with coronary syndrome
  Interventions: Other: Biological analysis of biomarkers
- 2 (Other): Subjects without coronary syndrome
  Interventions: Other: Biological analysis of biomarkers

INTERVENTIONS:
Other: Biological analysis of biomarkers — Biological analysis of biomarkers
  Arms: 1
Other: Biological analysis of biomarkers — Biological analysis of biomarkers
  Arms: 2

SUMMARY:
To assess diagnostic and prognostic value of new biomarkers in patients admitted for suspicion of non ST elevation acute coronary syndrome (NSTE ACS).

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years,
* subject about having a chest pain of coronary syndrome,
* subject about not having received heparin or LMWH

Exclusion Criteria:

* subject minor
* subject without informed consent,
* subject after receiving an anticoagulant treatment,
* transplanted heart, kidney or liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess diagnostic and prognostic value of new biomarkers in patients admitted for suspicion of non ST elevation acute coronary syndrome (NSTE ACS). | 24 months

SECONDARY OUTCOMES:
Compare the characteristics of biological markers to those of usual or innovative markers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis BONNET, MD, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone- Service cardiologie A, Marseille, France